CLINICAL TRIAL: NCT01109888
Title: Administration of Increased Dose of GnRH Antagonist for Coasting for Decreasing the Risk for Ovarian During Controlled Ovarian Stimulation(COH) for In Vitro Fertilisation(IVF)
Brief Title: Administration of Increased Dose of GnRH Antagonist for Coasting for Decreasing the Risk for Ovarian Hyperstimulation Syndrome( OHSS)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: there was no percipitant enrolled
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Levran D., M.D, IVF Unit, Wolfson Medical center
Other Study IDs: 12101967
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2010-04

CONDITIONS: Administration of Increased Dose of GnRH Antagonist for Coasting for Decreasing the Risk for Ovarian Hyperstimulation Syndrome( OHSS)
MeSH Terms: interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetrotide (Active Comparator)
  Interventions: Drug: Cetrotide

INTERVENTIONS:
Drug: Cetrotide

SUMMARY:
Coasting is one of the means to reduce the risk of OHSS for patients at risk for severe OHSS. During coasting gonadotrophin administration is withheld until serum E2 levels drop to a range considered safe. Prolonged coasting reduces the chance for implantation and pregnancy. The aim of the study is to explore whether an increased dose of GnRH Antagonist will shorten the coasting period without an adverse effect on cycle outcome.

DETAILED DESCRIPTION:
30 patients undergoing IVF using a GnRH antagonist protocol that present with a high response to gonadotrophin stimulation, will be randomized into one of two groups: group A - withdrawal of gonadotrophin support and continue a daily dose of 0.25 mg of the GnRH antagonist. group B - withdrawal of gonadotrophin support and continue a double daily dose of 0.5 mg of the GnRH antagonist.

The main outcome measures will be the duration of coasting (days)and the rate of serum E2 drop (%).

ELIGIBILITY:
Inclusion Criteria:30 women undergoing IVF cycle with GnRH Antagonist protocol under 35 years old.

E2 higher than 3000 pg/ml. -

Exclusion Criteria: 3 or more failed fresh IVF cycles.

-

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Enrollment: 0 (Actual)